CLINICAL TRIAL: NCT06535360
Title: Improving Efficacy and Safety of Pathogen Inactivation Strategies for Platelet Transfusion in Cardiac Surgical Patients on Cardiopulmonary Bypass
Brief Title: Efficacy of Pathogen Inactivation Strategies for Platelet Transfusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Magali Fontaine, Professor of Pathology, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00088613
Record Dates: First submitted 2024-05-06; First posted 2024-08-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Cardiopulmonary Bypass Surgery
MeSH Terms: interventions — Platelet Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRT PLTs stored in PAS (Experimental): FDA approved and already used in this patient population tested for non-inferiority
  Interventions: Biological: Platelet transfusion
- Non-PRT PLTs stored in platelet additive solution (PAS) (Active Comparator): FDA approved and already used in this patient population
  Interventions: Biological: Platelet transfusion

INTERVENTIONS:
Biological: Platelet transfusion — platelet administration through intravenous access

SUMMARY:
This is a prospective randomized clinical trial designed to determine the hemostatic ability of pathogen reduced platelet, when compared to non-pathogen reduced platelets suspended in platelet additive solution.

DETAILED DESCRIPTION:
The safety and efficacy of pathogen reduced (PRT) platelets (PLTs) have been investigated in several controlled clinical studies. Most of these clinical studies evaluated the efficacy of PRT PLTs during prophylactic transfusion evaluating post-transfusion platelet count increments, rather than platelet function during bleeding episodes. During massive transfusion events and immediate resuscitation, PLT transfusion is recognized as an important determinant of a positive patient outcome. PLT transfusion is important to control bleeding in patients undergoing cardiac surgery on cardiopulmonary bypass because cardiopulmonary bypass alters platelet function. Thus, transfusion of functional platelets is required to control bleeding post-operatively. In this context, the investigators propose to investigate whether efficient hemostasis associated with platelet transfusion differs with the use of pathogen reduced PRT PLTs compared to non-pathogen reduced PLTs that are suspended in platelet additive solution.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Preoperative evaluation for risk of transfusion: platelet count < 200,000/mcl, OR anticipated time on cardiopulmonary bypass > 90 min, OR complex cardiac surgery, OR use of preoperative antiplatelet therapy within 3-5 days of surgery.

Exclusion Criteria:

* Patient that lack the ability to consent
* Patients with the diagnosis of idiopathic thrombocytopenia purpura,
* Patient with the diagnosis of heparin-induced thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Maximum Amplitude (MA) of thromboelastography (TEG) | within 60 minutes including blood for TEG testing immediately pre transfusion and blood draw post transfusion
  ΔMA observed with platelet transfusion (difference in MA measured within an hour post transfusion to MA measured immediately pre-transfusion)

SECONDARY OUTCOMES:
Chest Tube Drainage | 24 hours
  The volume in ml of chest tube drainage during the first 24 hours post surgery
Red blood cell units Transfused | Within the first 24 Hrs Following Surgery
  number of red blood cell units transfused
Platelet Units Transfused | Within the first 24 Hrs Following Surgery
  number of platelet units transfused
Cryoprecipitate Units Transfused | Within the first 24 Hrs Following Surgery
  number of Cryoprecipitate Units Transfused
Plasma Units Transfused | Within the first 24 Hrs Following Surgery
  number of plasma units transfused

CONTACTS AND LOCATIONS:
Overall Officials: Magali Fontaine, MD, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No